CLINICAL TRIAL: NCT00889993
Title: Effect of Four Doses of Mixed Fiber on Satiety, Food Intake, Glucose, Insulin, and Gut Hormone Release
Brief Title: Satiety Response After Mixed Fiber Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 0701M00265
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Satiety
Keywords: Food intake; Gut hormones; Fiber; Visual analog scales

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Mixed Fiber Supplement — Breakfast Muffin containing 0g, 4g, 8g, and 12g of mixed fiber (total fiber amount as listed).

SUMMARY:
People who eat more dietary fiber have a lower body weight than people who eat less fiber. Potential mechanisms include greater feelings of satiety, reductions in food intake, changes in blood glucose, insulin, or gut hormones.

The investigators hypothesize that increasing doses of mixed fiber will influence satiety response, food intake, glucose, insulin, ghrelin, GLP-1, and PYY 3-36, in a dose-dependent manner, when given to subjects in muffins for breakfast.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* healthy men and women
* 18 and 65 years of age
* non-smoking
* not taking medications
* non-dieting (weight stable over last 3 months)
* BMI between 18 and 27
* able to give blood through an IV

Exclusion Criteria:

* irregular or erratic breakfast eating patterns
* food allergies to ingredients commonly found in muffins or pizza
* distaste for muffins or pizza
* BMI less than 18 or greater than 27
* weight change > 5 kg in last 3 months (intentional or unintentional)
* cardiovascular disease
* diabetes mellitus (fasting blood sugar > 126 mg/dl)
* cancer in prior 5 years (except basal cell carcinoma of skin)
* renal or hepatic disease
* Crohns disease
* ulcerative colitis
* any other gastrointestinal conditions that may affect digestion or absorption
* recent bacterial infection (< 3 months)
* chronic medication use
* history of drug or alcohol abuse in prior 6 months
* concurrent or recent intervention study participation
* vegetarians
* people who ate more than approximately 15 g of fiber per day
* pregnant or lactating women
* women with irregular menstrual cycles

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Satiety and Food Intake | November 2007 thru May 2008

SECONDARY OUTCOMES:
Glucose, Insulin, Gut Hormone Response | November 2007 thru October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota: General Clinical Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Willis HJ, Thomas W, Eldridge AL, Harkness L, Green H, Slavin JL. Glucose and insulin do not decrease in a dose-dependent manner after increasing doses of mixed fibers that are consumed in muffins for breakfast. Nutr Res. 2011 Jan;31(1):42-7. doi: 10.1016/j.nutres.2010.12.006. PMID 21310305